CLINICAL TRIAL: NCT04789590
Title: Determining the Effectiveness of the Geriatric Pain Measure ın Older Adults Attending a Gynecology Clinic
Brief Title: Multidimensional Geriatric Pain Assessment
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, AKİF BULUT, Principal Investigator, Uludag University
Other Study IDs: ABULUT
Record Dates: First submitted 2021-03-02; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Pain
Keywords: Geriatric Pain Measure; Pain Assessment; Elderly Adults
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This descriptive study was conducted on 100 patients who applied to the gynecology outpatient clinic to determine the effectiveness of the Geriatric Pain Measure (GPM) in elderly individuals. The data of the study were collected using the Patient Information Form, the GPM, and the Standardized Mini Mental State Examination (SMMSE). The mean GPM score of the elderly individuals, who had an average age of 70 (65-90), was found to be 27.37 (0-88), the sub-dimension mean scores were 9.52 (0-49.9), 7.14 (0-14.2), 4.76 (0-9.5), 2.38 (0-11.9), and 4.76 (0-11.9) respectively. It was determined that 54% of the patients had mild pain (0-29), 38% of them had moderate pain (30-69), and 8% of them had severe pain (70 and above). The findings of the present study were similar to the results of numerous other studies in which both the same scale and different scales were used to assess pain in elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older patients,
* Scoring 23 or above in the Standardized Mini Mental State Examination,
* Have no obstacle to answering questions,
* Not addicted to alcohol or other substances,
* No trauma in the last six months.

Exclusion Criteria:

* Patients younger than 65,
* Scoring less than 23 points in the Standardized Mini Mental State Examination,
* Who have a situation that prevents them from answering questions,
* Are addicted to alcohol or other substances,
* Trauma in the last six months.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Female patients 65 years of age or older who applied to gynecology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Determining the pain levels of patients aged 65 and over | 4 months
  The Geriatric Pain Measure is a 24-item multidimensional scale developed by Ferrell et al. (2000), for elderly individuals treated on an outpatient basis. Its validity and reliability in Turkish were confirmed by Dursun and Bektaş (2017). The Turkish version of the scale has five sub-dimensions: withdrawal due to pain (Factor 1; Items 19, 20, 22, 23); pain intensity (Factor 2; Items 1, 2, 3, 4, 5, 6); pain with movement (Factor 3; Items 9, 10, 11, 12); pain with strenuous activities (Factor 4; Items 7, 8, 18, 21, 24); and pain with other activities (Factor 5; Items 13, 14, 15, 16, 17). The total score is calculated by adding the "Yes" answers, and each item is multiplied by 2.38 and the total is converted into a score of between 0 and 100. Scores between 0 and 29 are considered to indicate mild pain, scores between 30 and 69 are considered to indicate moderate pain, and scores of 70 and above are considered to indicate severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: AKİF BULUT, Phd Student, Principal Investigator — Uludag University
Locations (1):
- Bursa Province Public Hospitals Union General Secretariat Health Sciences University Bursa High Specialization Education and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In the work permit obtained from Bursa Provincial Health Directorate, it was stipulated that the study data should not be shared.

REFERENCES:
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the Intensive Care Unit: executive summary. Am J Health Syst Pharm. 2013 Jan 1;70(1):53-8. doi: 10.1093/ajhp/70.1.53. PMID 23261901
- [Background] Blozik E, Stuck AE, Niemann S, Ferrell BA, Harari D, von Renteln-Kruse W, Gillmann G, Beck JC, Clough-Gorr KM. Geriatric Pain Measure short form: development and initial evaluation. J Am Geriatr Soc. 2007 Dec;55(12):2045-50. doi: 10.1111/j.1532-5415.2007.01474.x. Epub 2007 Nov 20. PMID 18031489
- [Background] Cavlak U, Yagci N, Bas Aslan U, Ekici G. A new tool measuring health-related quality of life (HRQOL): the effects of musculoskeletal pain in a group of older Turkish people. Arch Gerontol Geriatr. 2009 Sep-Oct;49(2):298-303. doi: 10.1016/j.archger.2008.11.002. Epub 2008 Dec 19. PMID 19101046
- [Background] Dahlhamer J, Lucas J, Zelaya C, Nahin R, Mackey S, DeBar L, Kerns R, Von Korff M, Porter L, Helmick C. Prevalence of Chronic Pain and High-Impact Chronic Pain Among Adults - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Sep 14;67(36):1001-1006. doi: 10.15585/mmwr.mm6736a2. PMID 30212442
- [Background] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Background] Hairi NN, Cumming RG, Blyth FM, Naganathan V. Chronic pain, impact of pain and pain severity with physical disability in older people--is there a gender difference? Maturitas. 2013 Jan;74(1):68-73. doi: 10.1016/j.maturitas.2012.10.001. Epub 2012 Oct 25. PMID 23103063
- [Background] Jackson T, Thomas S, Stabile V, Han X, Shotwell M, McQueen K. Prevalence of chronic pain in low-income and middle-income countries: a systematic review and meta-analysis. Lancet. 2015 Apr 27;385 Suppl 2:S10. doi: 10.1016/S0140-6736(15)60805-4. Epub 2015 Apr 26. PMID 26313056
- [Background] Zwakhalen SM, Hamers JP, Abu-Saad HH, Berger MP. Pain in elderly people with severe dementia: a systematic review of behavioural pain assessment tools. BMC Geriatr. 2006 Jan 27;6:3. doi: 10.1186/1471-2318-6-3. PMID 16441889
- [Background] Larsson C, Hansson EE, Sundquist K, Jakobsson U. Chronic pain in older adults: prevalence, incidence, and risk factors. Scand J Rheumatol. 2017 Jul;46(4):317-325. doi: 10.1080/03009742.2016.1218543. Epub 2016 Nov 25. PMID 27885914
- [Background] Layman Young J, Horton FM, Davidhizar R. Nursing attitudes and beliefs in pain assessment and management. J Adv Nurs. 2006 Feb;53(4):412-21. doi: 10.1111/j.1365-2648.2006.03735.x. PMID 16448484
- [Background] Sirsch E, Lukas A, Drebenstedt C, Gnass I, Laekeman M, Kopke K, Fischer T; Guideline workgroup (Schmerzassessment bei alteren Menschen in der vollstationaren Altenhilfe, AWMF Registry 145-001). Pain Assessment for Older Persons in Nursing Home Care: An Evidence-Based Practice Guideline. J Am Med Dir Assoc. 2020 Feb;21(2):149-163. doi: 10.1016/j.jamda.2019.08.002. Epub 2019 Oct 24. PMID 31668640
- [Result] Clough-Gorr KM, Blozik E, Gillmann G, Beck JC, Ferrell BA, Anders J, Harari D, Stuck AE. The self-administered 24-item geriatric pain measure (GPM-24-SA): psychometric properties in three European populations of community-dwelling older adults. Pain Med. 2008 Sep;9(6):695-709. doi: 10.1111/j.1526-4637.2008.00497.x. PMID 18816330
- [Result] Cornally N, McCarthy G. Chronic pain: the help-seeking behavior, attitudes, and beliefs of older adults living in the community. Pain Manag Nurs. 2011 Dec;12(4):206-17. doi: 10.1016/j.pmn.2010.12.006. Epub 2011 Feb 26. PMID 22117752
- [Result] Damico V, Murano L, Cazzaniga F, Dal Molin A. Pain prevalence, severity, assessment and management in hospitalized adult patients: a result of a multicenter cross sectional study. Ann Ist Super Sanita. 2018 Jul-Sep;54(3):194-200. doi: 10.4415/ANN_18_03_05. PMID 30284545
- [Result] Dursun G, Bektas H. Cultural Validation and Reliability of the Turkish Version of the Geriatric Pain Measure in the Elderly. Pain Pract. 2017 Apr;17(4):505-513. doi: 10.1111/papr.12473. Epub 2016 Jul 2. PMID 27370573
- [Result] Ferrell BA, Stein WM, Beck JC. The Geriatric Pain Measure: validity, reliability and factor analysis. J Am Geriatr Soc. 2000 Dec;48(12):1669-73. doi: 10.1111/j.1532-5415.2000.tb03881.x. PMID 11129760
- [Result] Horgas AL, Elliott AF, Marsiske M. Pain assessment in persons with dementia: relationship between self-report and behavioral observation. J Am Geriatr Soc. 2009 Jan;57(1):126-32. doi: 10.1111/j.1532-5415.2008.02071.x. Epub 2008 Nov 18. PMID 19054191
- [Result] Husebo BS, Strand LI, Moe-Nilssen R, Borgehusebo S, Aarsland D, Ljunggren AE. Who suffers most? Dementia and pain in nursing home patients: a cross-sectional study. J Am Med Dir Assoc. 2008 Jul;9(6):427-33. doi: 10.1016/j.jamda.2008.03.001. Epub 2008 Jun 2. PMID 18585645
- [Result] Iliffe S, Kharicha K, Carmaciu C, Harari D, Swift C, Gillman G, Stuck AE. The relationship between pain intensity and severity and depression in older people: exploratory study. BMC Fam Pract. 2009 Jul 28;10:54. doi: 10.1186/1471-2296-10-54. PMID 19638205
- [Result] Leong IY, Farrell MJ, Helme RD, Gibson SJ. The relationship between medical comorbidity and self-rated pain, mood disturbance, and function in older people with chronic pain. J Gerontol A Biol Sci Med Sci. 2007 May;62(5):550-5. doi: 10.1093/gerona/62.5.550. PMID 17522361
- [Result] Liberman O, Freud T, Peleg R, Keren A, Press Y. Chronic pain and geriatric syndromes in community-dwelling patients aged >/=65 years. J Pain Res. 2018 Jun 19;11:1171-1180. doi: 10.2147/JPR.S160847. eCollection 2018. PMID 29950889
- [Result] Motter FR, Hilmer SN, Paniz VMV. Pain and Inflammation Management in Older Adults: A Brazilian Consensus of Potentially Inappropriate Medication and Their Alternative Therapies. Front Pharmacol. 2019 Dec 2;10:1408. doi: 10.3389/fphar.2019.01408. eCollection 2019. PMID 31849664
- [Result] Nawai A, Leveille SG, Shmerling RH, van der Leeuw G, Bean JF. Pain severity and pharmacologic pain management among community-living older adults: the MOBILIZE Boston study. Aging Clin Exp Res. 2017 Dec;29(6):1139-1147. doi: 10.1007/s40520-016-0700-9. Epub 2017 Feb 21. PMID 28224474
- [Result] Park J, Cho B, Paek Y, Kwon H, Yoo S. Development of a pain assessment tool for the older adults in Korea: the validity and reliability of a Korean version of the geriatric pain measure (GPM-K). Arch Gerontol Geriatr. 2009 Sep-Oct;49(2):199-203. doi: 10.1016/j.archger.2008.07.010. Epub 2008 Sep 10. PMID 18786737
- [Result] Reynolds KS, Hanson LC, DeVellis RF, Henderson M, Steinhauser KE. Disparities in pain management between cognitively intact and cognitively impaired nursing home residents. J Pain Symptom Manage. 2008 Apr;35(4):388-96. doi: 10.1016/j.jpainsymman.2008.01.001. Epub 2008 Feb 15. PMID 18280101
- [Result] van Herk R, van Dijk M, Baar FP, Tibboel D, de Wit R. Observation scales for pain assessment in older adults with cognitive impairments or communication difficulties. Nurs Res. 2007 Jan-Feb;56(1):34-43. doi: 10.1097/00006199-200701000-00005. PMID 17179872
- [Result] Ware LJ, Epps CD, Herr K, Packard A. Evaluation of the Revised Faces Pain Scale, Verbal Descriptor Scale, Numeric Rating Scale, and Iowa Pain Thermometer in older minority adults. Pain Manag Nurs. 2006 Sep;7(3):117-25. doi: 10.1016/j.pmn.2006.06.005. PMID 16931417
- [Result] Woo J, Leung J, Lau E. Prevalence and correlates of musculoskeletal pain in Chinese elderly and the impact on 4-year physical function and quality of life. Public Health. 2009 Aug;123(8):549-56. doi: 10.1016/j.puhe.2009.07.006. Epub 2009 Aug 25. PMID 19709699

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-06-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT04789590/Prot_SAP_000.pdf
  • Informed Consent Form (2015-11-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT04789590/ICF_001.pdf